CLINICAL TRIAL: NCT03239054
Title: Prescribing Exercise as Medicine in Pregnancy: A Randomized Controlled Trial
Brief Title: Prescribing Exercise as Medicine in Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB issues
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Shilpa Babbar, MD, Principal Investigator, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 28028
Record Dates: First submitted 2017-07-23; First posted 2017-08-03 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Pregnancy
MeSH Terms: interventions — Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: participants will be randomized in a 1:1 fashion into the study group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Participants in the study group will complete the Parmed-X Pregnancy form and be provided with a prescription for exercise.
  Interventions: Behavioral: Physical activity
- Control Group (Other): The control group will be provided with the ACOG Pamphlet entitled "Exercise during pregnancy" and will be encouraged to become physically active during their pregnancy. They will receive routine care as scheduled.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Physical activity — pregnancy prescription for physical activity as part of prenatal care can increase healthy exercise behaviors during pregnancy
  Arms: Study Group
Behavioral: Control group — Information will be given as part of standard care
  Arms: Control Group

SUMMARY:
This study is a randomized controlled parallel arms trial. The purpose of this study is to evaluate if prescribing exercise in pregnancy can change maternal behavior towards exercise.

DETAILED DESCRIPTION:
This study is a randomized controlled parallel arms trial. The purpose of this study is to evaluate if prescribing exercise in pregnancy can change maternal behavior towards exercise. Once screened and consented, participants will be randomized to either the intervention or control group in a 1:1 fashion. The intervention group will receive the PARMED-X prescription and the control group will receive routine care as usual. Physical activity will be monitored with a Polar fitness tracking device.

Maternal and neonatal outcomes will be collected from the electronic medical record. Maternal outcomes include demographics, total gestational weight gain, pre-pregnancy body mass index (BMI), BMI at the time of delivery, mode of delivery, glucose screen value, presence or absence of gestational diabetes and presence or absence of hypertensive disorders of pregnancy. Neonatal outcomes include gestational age at delivery, birth weight, Apgar scores, arterial cord blood gases.

Psychological outcomes will also be assessed using several validated scales in pregnancy including The Edinburgh Postnatal Depression Scale (EPDS) and The State Trait Anxiety Inventory (STAI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years of age
* Singleton pregnancy
* Gestational age at or less than 20 0/7 weeks at the time of enrollment
* Low risk pregnancy
* Willing and able to participate in a more active lifestyle/exercise program
* Smart phone able to add the "Flow mobile app".

Exclusion Criteria:

* Twins or higher order multiple gestations
* Known congenital anomaly
* Underweight BMI ( BMI less than 18.50)
* High risk pregnancy - ie. hypertension, pre-existing diabetes
* Women with a known contraindication to exercise
* Persistent 2nd or 3rd trimester vaginal bleeding
* Hemodynamically significant heart disease
* Restrictive lung disease
* Incompetent cervix or cerclage
* Placenta previa
* Premature labor or rupture of membranes
* Preeclampsia
* Severe anemia
* Poorly controlled hypertension, seizure disorder, or hyperthyroidism
* Known intrauterine growth restriction
* Not cleared for exercise by the "Contraindications to Exercise from PARMED-X" form
* PAVS score greater than or equal to 150 minutes/week

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
PARmed-X: Change in number of steps (physical activity level) | 1 year
  change in number of steps (physical activity level)

SECONDARY OUTCOMES:
PARMed-X: Gestational Weight Gain | 1 year
  Gestational Weight Gain

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Babbar, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No